CLINICAL TRIAL: NCT01496300
Title: Randomised Controlled Double-blind Monocenter Therapy Study Validating the Benefit From Information Provided by Image Free Navigation System on the Precision of the Placement of Acetabular Component in Patients Undergoing Primary THA
Brief Title: Benefit of Orthopedic Navigation in the ARThroplasty of the Hip
Acronym: BONARTH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAG-G-H-1103
Record Dates: First submitted 2011-12-15; First posted 2011-12-21 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Osteoarthritis, Hip; Arthritis, Rheumatoid; Femur Head Necrosis
Keywords: Navigation OrthoPilot Hip TEP THA
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis, Rheumatoid; Femur Head Necrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual (Sham Comparator): Manual Implantation of THA
  Interventions: Procedure: Manual Intervention
- Navigated (Experimental): Navigated Implantation of THA
  Interventions: Procedure: Navigated Intervention

INTERVENTIONS:
Procedure: Manual Intervention — Implantation of acetabular component without the use of the navigation system information
  Other Names: Conventional THA
  Arms: Manual
Procedure: Navigated Intervention — Navigated implantation of acetabular component using OrthoPilot image free navigation system
  Other Names: Computer assisted orthopedic surgery
  Arms: Navigated

SUMMARY:
This study was initiated to investigate the impact of the computer based image free navigation on the precision of the cup implantation. The implantation of the acetabular component (cup) is known to be a critical step in hip endoprosthetics. The cup position influences significantly the function, the absence of pain and the longevity of the artificial hip joint. The image free navigation system OrthoPilot is used to control the positioning of the cup during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Indication for primary cementless total hip endoprosthesis implantation with Bicontact stem and Plasmacup
* Diagnoses: primary or secondary coxarthrosis, rheumatoid arthritis, femoral head necrosis
* Age ≥ 50 Years
* ASA score <4
* Patient signed the informed consent

Exclusion Criteria:

* Excessive damage to the hip joint (e.g. dysplasia)
* Severe deformities of the pelvis, femoral bone or knee
* Unfeasibility of landmark palpation (e.g. due to adiposity)
* Acute or chronic infection
* Pregnancy
* Patients not available for follow-up-examination at the center
* Patients exceeding 10 mSv effective radiation dose because of previous scientific or clinical exposition during the past 10 years

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of improvement of the implantation accuracy of acetabular component by navigation compared to manual implantation | 3 months
  The ratio of implantations within the intraoperatively adjusted safe zone of Lewinnek (target anteversion +/-10°, target inclination +/-10°), proved by a CT-scan control measurement.

SECONDARY OUTCOMES:
Comparison of implantation precision, postoperative function and complication rates with vs. without gaining information from navigation system. | 3 months
  The ratio of implantations within the intraoperatively determined safe zone of 5° (target anteversion +/-5°, target inclination +/- 5°) Geometric deviation from the target implantation position Range of Motion Harris hip score 3 months postoperative Complication rate until 3 months Correlation of manual and ultrasound registration of the anterior pelvic plane (independent from therapy group) Proposal and validation of a combined Hip Alignment Score for navigated implantation

CONTACTS AND LOCATIONS:
Overall Officials: Hartmuth Kiefer, Prof. Dr., Principal Investigator — Lukas Krankenhaus Bünde
Locations (1):
- Lukas-Krankenhaus, Bünde, Germany